CLINICAL TRIAL: NCT06841796
Title: The Young Men's Christian Association (YMCA) Healthy Lifestyle Program for Prediabetes
Brief Title: The YMCA Healthy Lifestyle Program for Prediabetes
Acronym: Y-HELP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Young Men's Christian Association of the Blue Water Area (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Sushma Reddy, MD, Principal Investigator, Young Men's Christian Association of the Blue Water Area
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIS-2024-173
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: PreDiabetes
Keywords: prediabetes; diabetes prevention; prevention of type 2 diabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Randomized controlled 24 week single center in-person trial
Who Masked: Outcomes Assessor
Masking Description: All study personnel will be blinded to the "blinded' CGM data until the participant completes all study visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 : Intervention with Stelo (Active Comparator): Stelo CGM
  Interventions: Device: Real time continuous glucose monitor (Stelo)
- Group 2 : control (No Intervention): Group 2 will only wear a blinded CGM for 10 days at 6,12 and 24 weeks

INTERVENTIONS:
Device: Real time continuous glucose monitor (Stelo) — Real time CGM will be worn continuously for 24 weeks. Participants will be able to see the glucose data from the CGM facilitating changes in nutritional habits and physical activity
  Arms: Group 1 : Intervention with Stelo

SUMMARY:
The goal of this 26 week randomized controlled clinical trial is to learn if using a real time continuous glucose monitor (CGM) in a healthy lifestyle program for adults with prediabetes at the YMCA can improve glucose levels, dietary habits and physical activity The main questions it aims to answer is

* Does use of a CGM improve the percent of time spent with glucose values between 70-140 mg/dl
* Does use of a CGM improve nutritional habits as measured by Picture Your Plate (PYP) score
* Does use of a CGM improve physical activity as measured by International Physical Activity Questionnaire (IPAQ) score

Researchers will compare individuals using real time CGM to those not using CGM

Participants will be asked to:

* attend weekly health coach sessions for 12 weeks followed by 3 monthly sessions.
* attend a YMCA class of their choice
* fill out questionnaires at baseline, 12 and 24 weeks
* have an A1c blood test at baseline, 12 and 24 weeks.
* wear a CGM.

All participants will wear a blinded CGM at baseline. The intervention group will wear a real time CGM for 24 weeks. The control group will wear a blinded CGM for 10 days at 6, 12 and 24 weeks

DETAILED DESCRIPTION:
BACKGROUND:

Diabetes has a significant impact on physical, social and mental well-being and causes significant morbidity and mortality in the United States. The total direct estimated costs of diagnosed diabetes have increased from $227 billion in 2012 to $307 billion in 2022.

In 2021, 38.1 million adults aged 18 years or older (14.7% of all US adults) had diabetes with a higher prevalence of 29.2% among those aged 65 years or older. An estimated 97.6 million adults had prediabetes in 2021.

The Diabetes Prevention Program (DPP) study published in 2002 clearly showed the benefit of lifestyle intervention in reducing the risk of developing type 2 diabetes by 58% compared to placebo. The Program worked particularly well for participants ages 60 and older, lowering their chances of developing type 2 diabetes by 71 percent. However, the retention rate for the DPP program has been 32% at 10 months with only 17% achieving all three goals of weight loss, physical activity ≥ 150 min per week and low fat diet. In fact, over the 20 years since the study was published, the incidence and prevalence of diabetes have dramatically increased with prediabetes affecting more than one third of the adult population. It is clear that a new approach is needed to prevent individuals with prediabetes progressing to diabetes

RATIONALE:

CGM has been shown to be an effective behavior modification tool in individuals with diabetes resulting in improvement in A1c and weight loss. Individuals with diabetes wearing a CGM were more likely to modify their physical activity and eating habits based on the real time glucose levels from the CGM.

The Diabetes Prevention Program (DPP) has been successfully implemented in the YMCA setting using health coaches and a modified curriculum. However, overall enrollment in Diabetes Prevention Programs is low with only 16% (351/2200) of those contacted attending an information session and only 11.3% (228) enrolling in the YMCA DPP and persisting through week 9. Overall retention rate for DPP at University of Michigan was 63% of participants through 18 weeks and 32% of participants through 44 weeks.

It was felt that a healthy lifestyle program led by a YMCA health coach incorporating the real time feedback of glucose data from the CGM and elements of the DPP curriculum could effectively help individuals with prediabetes make the necessary lifestyle changes to prevent diabetes.

PRIMARY OBJECTIVE:

To determine if a healthy lifestyle program at the YMCA incorporating CGM in individuals with prediabetes can improve glucose levels, dietary habits and physical activity

SECONDARY OBJECTIVE:

To determine if a healthy lifestyle program at the YMCA incorporating CGM in individuals with prediabetes can have a beneficial effect on weight, body mass index (BMI), waist circumference, body fat percentage, self-perceived health/wellness and participant satisfaction

STUDY DESIGN:

This is a randomized controlled single center 24 week in-person trial intended to investigate the effect of CGM in improving glucose levels, physical activity and nutritional habits in individuals with prediabetes in a YMCA Healthy Lifestyle Program.

In this trial, 84 participants with prediabetes will be randomly assigned 1:1 to two groups. Baseline A1c and BMI will be taken into account during randomization to ensure that the two groups are similar.

All participants will undergo baseline assessment including wearing a blinded CGM for 10 days. The intervention arm (Group 1) will wear real time CGM continuously for 24 weeks and the control arm (Group 2) will wear only a blinded CGM at week 6, 12 and 24.

Both groups will attend sessions with a health coach weekly for the first 12 weeks followed by 3 monthly sessions. These sessions will include physical fitness activities and educational information on nutrition, motivation, coping, stress management and glucose levels.

A1c, glucose management indicator (GMI), nutritional, physical, diabetes empowerment scale modified for prediabetes (DES) and self-perceived health/wellness assessments will be obtained at baseline, 12 and 24 weeks. Weight, BMI, waist circumference and body fat percentage measurements will be obtained at baseline, 4, 8, 12, 16, 20 and 24 weeks. Semi-structured interviews will be performed on a cross section of participants about their attitudes and perceptions with CGM usage and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* ● Adults 18 years or older AND

  * A diagnosis of prediabetes as defined by:

    * Fasting glucose 100-125 mg/dl OR
    * A1c 5.7-6.4%

Exclusion Criteria:

* Pregnancy
* Previous CGM use
* Lack of smart phone/smart device
* Use of steroids
* Active cancer treatment
* Active chronic infection requiring long term use of antibiotics
* Terminal illness
* Dementia, mental impairment
* Non English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time in tight range (TITR) | Assessed at baseline, 6,12 and 24 weeks
  Percent of time with glucose values in the range of 70-140 mg/dl
PYP | Assessed at baseline, 12 and 24 weeks
  Change in picture your plate (PYP) score. The score ranges from 0 to 96 with a higher score indicating a healthier diet. A score < 40 indicates greater likelihood of an unhealthy dietary pattern with much room for improvement. A PYP score greater than 60 indicates a healthful dietary pattern, although there may be some specific eating behaviors that could be improved.
IPAQ | Assessed at baseline, 12 and 24 weeks
  Change in International Physical Activity Questionnaire (IPAQ) score. This score is reported as Metabolic Equivalent (MET) minutes/week. Values can range from 0 to 4000 with a higher value indicating more physical activity

SECONDARY OUTCOMES:
A1c | baseline, 12 and 24 weeks
  Change in point-of-care A1c results
Change in BMI | baseline, 4,8,12,16,20 and 24 weeks
  Assessed by Tanita scale through measurements of height and weight. BMI is reported as kg/m2
Change in weight | baseline, 4,8,12,16,20 and 24 weeks
  Assessed by Tanita scale. Measured in pounds
Change in waist circumference | baseline, 4,8,12,16,20 and 24 weeks
  Assessed by Tanita scale. Measured in inches
Change in body fat percentage | baseline, 4,8,12,16,20 and 24 weeks
  Assessed by Tanita scale. Measured as body fat percentage

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Reddy, MD, Principal Investigator — Young Men's Christian Association of the Blue Water Area; Annette Gilmer, MD, MPH, Principal Investigator — Young Men's Christian Association of the Blue Water Area
Locations (1):
- YMCA of the Blue Water Area, Port Huron, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers

DOCUMENTS (1):
  • Informed Consent Form (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT06841796/ICF_000.pdf